CLINICAL TRIAL: NCT07090486
Title: Impact of Nirmatrelvir-ritonavir on Changes in Healthcare Utilization and Frailty Following COVID-19: a Difference-in-difference Analysis
Brief Title: A Study to Understand How the Use of Paxlovid Affected Healthcare Use in People With Pre-existing Conditions.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4671067
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
Keywords: Coronavirus-19 disease (COVID-19); Kaiser Permanente Southern California (KPSC); post-COVID conditions (PCC); Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2); Long COVID; nirmatrelvir-ritonavir
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants who received nirmatrelvir-ritonavir: Patients with cardio-pulmonary conditions
  Interventions: Drug: nirmatrelvir-ritonavir
- Participants who did not received nirmatrelvir-ritonavir: Patients with cardio-pulmonary conditions

INTERVENTIONS:
Drug: nirmatrelvir-ritonavir — Paxlovid standard of treatment care
  Other Names: Paxlovid
  Groups: Participants who received nirmatrelvir-ritonavir

SUMMARY:
This is a cohort study that will include Paxlovid (nirmatrelvir-ritonavir) treatment eligible for people with a positive SARS-CoV-2 diagnostic test and at least one COVID-19 symptom. This study will look at the change in Post Covid Conditions measured by the number of outpatients, Emergency department, urgent care and inpatient visits before and after COVID-19 between those who did and did not receive Paxlovid. In addition, changes in frailty post-acute infection will be evaluated, in a separate analysis. It is hypothesized that individuals with COVID-19 who received Paxlovid will have a smaller post-COVID-19 increase (vs pre-COVID) in PCC healthcare utilization (i.e., cardiopulmonary) in comparison to patients with COVID-19 who did not receive Paxlovid.

ELIGIBILITY:
Inclusion Criteria:

* Developed at least one COVID-19 symptom between Apr 1, 2022 through Dec 31, 2023
* A positive lab-confirmed polymerase chain reaction (PCR) SARS-COV-2 test 5 days after symptom onset (primary analysis).
* Continuous enrollment in KPSC health plans for at least 1 year (allowing for a 31-day gap to account for potential delays in membership renewal) before the date of symptom onset
* Active membership in KPSC health plans for at least 31 days after the date of symptom onset
* Eligible for nirmatrelvir-ritonavir defined by age and CDC-defined risk factors for severe COVID-19

Exclusion Criteria:

* Individuals on another medication that is contraindicated for treatment with nirmatrelvir-ritonavir defined as having any prescription drug claim in the 90 days prior to COVID-19 symptom onset
* Receipt of any COVID-19 antiviral (molnupiravir, remdesivir, nirmatrelvir/ritonavir) or monoclonal antibody treatment (bamlanivimab, bebtelovimab, casirivimab/imdevimab, cilgavimab/tixagevimab, otrovimab,) <180 days prior to COVID-19 symptom onset
* Any positive SARS-CoV-2 test, including self-reported tests, <180 days prior to COVID-19 symptom onset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Members of the Kaiser Permanente Southern California integrated healthcare delivery system.
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Cardio-pulmonary Measurement A: Change in rate of cardiopulmonary-related healthcare utilization in patients that received nirmatrelvir-ritonavir compared to not received. | 180 days before COVID-19 symptoms to 180 days after or 365 days after

SECONDARY OUTCOMES:
Frailty Measurement A: Change in frailty measured by Frailty score Median (IQR) in patients that did receive in patients nirmatrelvir-ritonavir compared to not received. | During Pre-period: 12 months prior to symptom onset Frailty score Median (IQR) to 12 months after.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671067